CLINICAL TRIAL: NCT00350168
Title: An 8-week Multicenter Study to Evaluate the Efficacy and Safety of Orally Administered Valsartan/Amlodipine Combination Based Therapy Versus Amlodipine Monotherapy in Patients With Stage II Hypertension
Brief Title: Efficacy & Safety of Orally Administered Valsartan/Amlodipine Combo Therapy vs Amlodipine Monotherapy in Patients With Stage II Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2403
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Blood pressure; Venous pressure; Systolic pressure; Diastolic pressure; Pulse pressure
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination

INTERVENTIONS:
Drug: valsartan + amlodipine

SUMMARY:
The purpose of this study is to evaluate the blood pressure lowering effects of a valsartan/amlodipine combination treatment and amlodipine monotherapy for the treatment of stage II hypertensive patients (MSSBP ≥ 160 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Moderate to severe high blood pressure. This is defined as a systolic pressure (the top number) greater than or equal to 160 mmHg and less than 200 mmHg.

Exclusion Criteria:

* History of allergy or hypersensitivity to ARBs, CCBs, thiazide diuretics
* Inability to stop all prior blood pressure medications safely
* Systolic BP ≥ 200 mmHg and/or diastolic BP ≥ 120 mmHg
* Controlled blood pressure (systolic BP < 140 mmHg) taking more than 3 antihypertensive medications at screening
* Systolic BP ≥ 140 mmHg and < 180 mmHg taking more than two antihypertensive medications at screening
* Systolic BP ≥ 180 mmHg taking more than one antihypertensive medication at screening
* History of stroke, angioplasty, coronary artery bypass graft surgery, heart attack or unstable angina
* Type 1 diabetes
* Poorly controlled Type 2 diabetes
* History of heart failure
* Arrhythmia
* Significant valvular heart disease
* Active gout
* History of autoimmune diseases
* History of multiple drug allergies
* Liver disease
* Pancreatic injury within 1 year of screening
* Evidence of kidney impairment or history of dialysis
* Any surgical or medical condition which might alter the absorption, distribution, metabolism, or excretion of any drug. This could include currently active gastritis, ulcers, or gastrointestinal/rectal bleeding, or urinary tract obstruction.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, would be excluded UNLESS they are post-menopausal, surgically sterile OR are using acceptable methods of contraception. The use of hormonal contraceptives is not allowed
* Pregnant or nursing (lactating) women
* History of malignancy of any organ system within the past five years
* Any severe, life-threatening disease within the past five years
* History of drug or alcohol abuse within the last 2 years.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MSSBP at week 4

SECONDARY OUTCOMES:
Change from baseline MSSBP after 2 and 8 weeks of treatment
Change from baseline MSDBP after 2, 4 and 8 weeks of treatment
Proportion of patients reaching overall BP control (MSSBP < 140 mmHg and MSDBP < 90mmHg) after 8 weeks of treatment
Evaluation of safety and tolerability after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals Corp, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Destro M, Luckow A, Samson M, Kandra A, Brunel P. Efficacy and safety of amlodipine/valsartan compared with amlodipine monotherapy in patients with stage 2 hypertension: a randomized, double-blind, multicenter study: the EX-EFFeCTS Study. J Am Soc Hypertens. 2008 Jul-Aug;2(4):294-302. doi: 10.1016/j.jash.2008.01.004. Epub 2008 Jun 2. PMID 20409909